CLINICAL TRIAL: NCT05730543
Title: Ethnic Lip Augmentation With Hyaluronic Acid Filler: Utilization of a Validated Lip Fullness Scale and Determining Pre Injection Lips Size Preference and Post Injection Patient Satisfaction
Brief Title: Ethnic Lip Augmentation With Hyaluronic Acid Filler
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DeNova Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIPS-DAYAN-22
Record Dates: First submitted 2022-12-01; First posted 2023-02-16 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Lip Augmentation; Lip Fullness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Volbella or Juvederm Ultra XC filler (Experimental): Injection will not exceed a total of 4 cc of hyaluronic acid filler for combined treatment sessions (initial treatment + possible touch up treatment session).
  Interventions: Drug: Volbella or Juvederm Ultra XC filler

INTERVENTIONS:
Drug: Volbella or Juvederm Ultra XC filler — Hyaluronic acid filler

SUMMARY:
Lip augmentation using hyaluronic acid filler in females with Fitzpatrick skin type V-VI

DETAILED DESCRIPTION:
Using the revised Allergan Lip Fullness Scale (LFS) to improve post injection patient satisfaction in women with Fitzpatrick skin type (FPST) 5 and 6 (examples: Hispanic, African descendants, Indigenous Australians).

ELIGIBILITY:
Inclusion Criteria:

1. Females age 21 and above, with FPST 5 or 6, undergoing lip filler augmentation
2. Subjects will be required not to have had previous lip filler, fat injections, or other lip treatments in the last 12 months.
3. Subjects that understand the purpose and aspects of the study, freely sign the informed consent, complete the required treatment and follow up protocol.

Exclusion Criteria:

1. Females below the age of 21
2. Male patients
3. Subjects with LFS 5
4. Fitzpatrick skin Type 1-4
5. Subjects who have had previous lip filler, fat injections or other surgical lip augmentation in the last 12 months
6. Subjects who are pregnant or nursing
7. Subjects with a known allergy or sensitivity to any component of the study ingredients.
8. Subjects that do not understand the purpose and aspects of the study, do not sign the consent, and do not complete the required treatment and follow up visit will also be excluded.
9. Subjects with a history of bleeding disorders (Vitamin K deficiency, liver disease, renal disease, iatrogenic or otherwise). This includes persons who have undergone therapy with thrombolytics, anticoagulants, or inhibitors of platelet aggregation in the preceding 3 weeks (such as Coumadin, Plavix, heparin analogues)
10. Subjects should not be taking aspirin, nonsteroidal anti-inflammatory medications, St. John's Wort, or high doses of Vitamin E supplements within 7 days prior to the start of the study
11. Subjects with active inflammation or infection in the area of treatment

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Lip size | 1 month
  The size of lip most desired based on the LFS scale. The possible choices are: 1) Minimal: flat or nearly flat contour, minimal red lip show. 2) Mild: some red lip show, no lower lip pout. 3) Moderate: Moderate red lip show with slight lower lip pout. 4) Marked: significant red lip show and lower lip pout, upper lip with moderate pout. 5) Very Marked: very significant red lip show, significant upper and lower lip pout.
Satisfaction level | 1 month
  Satisfaction levels relative to baseline via the FACE-Q questionnaire. The questionnaire asks the following questions: 1) The shape of your lower lip? 2) How well your lips suit your face? 3) How nice your lips look when you smile. 4) How full your lower lip looks? 5) The style of your lips (e.g. pouty, natural)? 6) The shape of your upper lip? 7) How turned up your upper lip (cupids bow) looks? 8) The size of your lips? 9) How the outer corners of your lips look when your face is relaxed (still)? 10) How full your lips look? The possible choices for each question are as follows: very dissatisfied (1), somewhat dissatisfied (2), somewhat satisfied (3), very satisfied (4). Responses of very satisfied signify a more positive outcome. Overall scores closer to 40 signify a more favorable satisfaction level.

SECONDARY OUTCOMES:
LFS by age group | 1 month
  LFS preference by age group (21-40 years old vs. 41+ years old). The size of lip most desired based on the LFS scale. The possible choices are: 1) Minimal: flat or nearly flat contour, minimal red lip show. 2) Mild: some red lip show, no lower lip pout. 3) Moderate: Moderate red lip show with slight lower lip pout. 4) Marked: significant red lip show and lower lip pout, upper lip with moderate pout. 5) Very Marked: very significant red lip show, significant upper and lower lip pout.
Improvement level | 1 month
  Subjects will determine which LFS scale category they would like to be and then based upon final visit they will rate themselves again as to where they actually fall on the scale. Investigator will do the same but only at final visit.

CONTACTS AND LOCATIONS:
Locations (1):
- DeNova Research, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Private study

REFERENCES:
- [Result] Dayan SH, Bacos JT, Gandhi ND, Ho TT, Kalbag A. Assessment of the Impact of Perioral Rejuvenation With Hyaluronic Acid Filler on Projected First Impressions and Mood Perceptions. Dermatol Surg. 2019 Jan;45(1):99-107. doi: 10.1097/DSS.0000000000001613. PMID 30059389
- [Result] Werschler WP, Fagien S, Thomas J, Paradkar-Mitragotri D, Rotunda A, Beddingfield FC 3rd. Development and validation of a photographic scale for assessment of lip fullness. Aesthet Surg J. 2015 Mar;35(3):294-307. doi: 10.1093/asj/sju025. PMID 25805282
- [Result] Burgess C, Awosika O. Ethnic and Gender Considerations in the Use of Facial Injectables: African-American Patients. Plast Reconstr Surg. 2015 Nov;136(5 Suppl):28S-31S. doi: 10.1097/PRS.0000000000001813. PMID 26441107